CLINICAL TRIAL: NCT06950853
Title: ESCAPE : Evaluation of Spinal Conservation by Endoscopic Procedures to Avoid Fusion
Acronym: ESCAPE
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Other Study IDs: CHUBX 2023/60
Record Dates: First submitted 2025-04-22; First posted 2025-04-30 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Spinal Stenosis; Spondylolisthesis
Keywords: spine; care; surgery
MeSH Terms: conditions — Spinal Stenosis; Spondylolisthesis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The recent development and expansion of endoscopic surgery has made it possible to offer an alternative to this therapeutic escalation. This method allows decompression procedures to be performed using optimized and minimally destructive surgical approaches, which contributes to preserving the physiological function of the lumbar spine and in particular its stability.

The main hypothesis of the research is that the use of endoscopic techniques for decompression of the lumbar spine allows a reduction in the indication for lumbar arthrodesis.

ELIGIBILITY:
Inclusion Criteria:

* Patient ≥ 18 years old
* Patient consulting for a medical reason involving a spinal pathology in the investigating center :

Syndrome adjacent to an old lumbar arthrodesis defined on preoperative radiographs by an antero-posterior translation > 3 mm, segmental kyphosis > 10° or a disc height reduced by more than 50%, or on preoperative MRI by central stenosis of grade C or D of the Schizas classification or a herniated disc Grade 1 or 2 degenerative spondylolisthesis, i.e. with slippage less than 50% of the depth of the underlying vertebral body.

Lumbar stenosis complicating lumbar scoliosis defined by a deformation with rotation of the vertebral bodies on a frontal radiograph (absence of centering of the spinous process between the two pedicles of the vertebra concerned) and a Cobb angle greater than 20° or a rotational dislocation .

- Indication for spinal surgery by endoscopy

Exclusion Criteria:

* Patient under guardianship or curatorship,
* Persons deprived of liberty by judicial or administrative decision,
* Persons undergoing psychiatric treatment under duress requiring the consent of the legal representative
* Persons unable to express their consent,
* Persons under legal protection,
* Patient not affiliated to a social protection scheme.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: lumbar spine surgery patients with pathologies eligible for arthrodesis surgery
Sampling Method: Non-Probability Sample
Enrollment: 375 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2027-08-01 (Estimated); Study Completion 2028-08-13 (Estimated)

PRIMARY OUTCOMES:
Surgical reintervention | one year
  rate of surgical reinterventions within the year for arthrodesis of the operated segment.

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin BOUYER, PROF, Principal Investigator — University Hospital, Bordeaux
Locations (10):
- France (10):
  - Hôpital Pellegrin, Centre Hospitalier Universitaire de Bordeaux, Bordeaux
  - Clinique du dos de Bordeaux -Terrefort, Bruges
  - CHU Lille, Lille
  - Centre orthopédique SANTY, Lyon
  - Hôpital CLAIRVAL, Marseille
  - CH de Narbonne, Narbonne
  - Centre hospitalier Privé Sainte Marie, Osny
  - Clinique du sport, Pessac
  - Institut locomoteur de l'Ouest-Rachi, Saint-Grégoire
  - Cabinet Orthosud Montpellier-Clinique Saint Jean, Saint-Jean-de-Védas

IPD SHARING:
Plan to Share IPD: No